CLINICAL TRIAL: NCT01096914
Title: Radiofrequency Ablation Versus Laser Ablation for the Treatment of Small Hepatocellular Carcinoma: a Randomized Controlled Trial
Brief Title: Radiofrequency Versus Laser Ablation for Hepatocellular Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardarelli Hospital (Other)
Responsible Party: Principal Investigator, Giovan Giuseppe Di Costanzo, MD, Cardarelli Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: epatologia1
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Carcinoma, Hepatocellular; Neoplasms, Liver
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiofrequency (Active Comparator): patients treated with percutaneous radiofrequency ablation
  Interventions: Procedure: percutaneous radiofrequency ablation
- laser (Active Comparator): Patients treated with percutaneous laser ablation
  Interventions: Procedure: percutaneous laser ablation

INTERVENTIONS:
Procedure: percutaneous radiofrequency ablation — Procedure: Radiofrequency ablation For RFA, we used a commercially available system (Valleylab, Tyco Healthcare, Boulder, CO, USA) and a 17-gauge "cool-tip" needle electrode with a 3cm exposed tip. The needle is inserted percutaneously under ultrasound guidance in the HCC nodule and treatment lasts 12 minutes. For nodules larger than 3cm in diameter, 2 insertions are used. In a period of six months, treatment may be repeated for no more than three times. When, after treatment, CT or MRI show a residual nodule activity of 10% or less, percutaneous ethanol injection may be done. If the residual activity is of 50% or more transarterial chemoembolization may be used.
  Other Names: Cool-tip ablation system - Valleylab, USA
  Arms: Radiofrequency
Procedure: percutaneous laser ablation — Procedure: Laser ablation For LA, we used a commercially available system (Echolaser XVG system, Esaote El.En., Florence, Italy) and four optical fibers,inserted into the cancer through four 21-gauge needles. The treatment lasts 6 minutes. For nodules larger than 3 cm in diameter, two treatments are done. In a period of six months, treatment may be repeated for no more than three times. When, after treatment, CT or MRI show a residual nodule activity of 10% or less, percutaneous ethanol injection may be done. If the residual activity is of 50% or more transarterial chemoembolization may be used.
  Other Names: Echolaser XVG system, Italy
  Arms: laser

SUMMARY:
The purpose of this study is to prospectively compare percutaneous radiofrequency ablation (RFA) versus percutaneous laser ablation (LA) for the treatment of small hepatocellular carcinoma in patients with cirrhosis.

DETAILED DESCRIPTION:
Percutaneous ablation is a safe and effective therapy for cirrhotic patients with HCC when resection or liver transplantation is not possible. Among the various percutaneous local ablative therapies, radiofrequency ablation (RFA) has attracted the greatest interest because of its effectiveness and safety for single HCC ≤ 5.0cm or ≤3 HCC nodules ≤3cm. Some studies have shown that laser ablation (LA) may be as effective as RFA in the treatment of HCC. However, RFA and LA are different techniques and, in different cases (for example: size or site of HCC nodule), each of these procedures may have some advantages or disadvantages. Therefore there is the need for a prospective randomized controlled study to compare RFA and LA in patients with small HCC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable HCC or who refused surgery
* A solitary HCC ≤ 5.0cm in diameter, or multiple HCC ≤ 3 lesions, each ≤ 3.0cm in diameter
* Child-Pugh class A or B
* Platelet count correctable to > 40,000/mm3, INR correctable to < 2.0
* No previous treatment of HCC

Exclusion Criteria:

* Other severe concomitant diseases that may reduce life expectancy
* History of encephalopathy, refractory ascites or variceal bleeding
* Vascular invasion or extrahepatic metastasis
* Human immunodeficiency virus (HIV) infection
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2009-01; Primary Completion 2012-09 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Tumor response | four weeks after treatment
  Complete ablation of the HCC nodule, defined as absence of contrast enhancement of the nodule at CT or MRI imaging

SECONDARY OUTCOMES:
overall survival | 12 months after last treatment
  Time from randomization to death. Patients alive at the end of follow-up are censored.
time to local recurrence | 12 months after treatment
  the time from complete tumor ablation to reappearance of arterial enhancement on CT or MRI either within a treated tumor or near its borders

CONTACTS AND LOCATIONS:
Overall Officials: Giovan Giuseppe Di Costanzo, MD, Principal Investigator — Liver Unit - Cardarelli Hospital - Via A Cardarelli 9 - 80131 Naples-Italy
Locations (1):
- Liver Unit - Cardarelli Hospital, Naples, Italy

REFERENCES:
- [Background] Pacella CM, Francica G, Di Lascio FM, Arienti V, Antico E, Caspani B, Magnolfi F, Megna AS, Pretolani S, Regine R, Sponza M, Stasi R. Long-term outcome of cirrhotic patients with early hepatocellular carcinoma treated with ultrasound-guided percutaneous laser ablation: a retrospective analysis. J Clin Oncol. 2009 Jun 1;27(16):2615-21. doi: 10.1200/JCO.2008.19.0082. Epub 2009 Mar 30. PMID 19332729
- [Background] Germani G, Pleguezuelo M, Gurusamy K, Meyer T, Isgro G, Burroughs AK. Clinical outcomes of radiofrequency ablation, percutaneous alcohol and acetic acid injection for hepatocelullar carcinoma: a meta-analysis. J Hepatol. 2010 Mar;52(3):380-8. doi: 10.1016/j.jhep.2009.12.004. Epub 2010 Jan 17. PMID 20149473
- [Background] Ferrari FS, Megliola A, Scorzelli A, Stella A, Vigni F, Drudi FM, Venezia D. Treatment of small HCC through radiofrequency ablation and laser ablation. Comparison of techniques and long-term results. Radiol Med. 2007 Apr;112(3):377-93. doi: 10.1007/s11547-007-0148-2. Epub 2007 Apr 20. English, Italian. PMID 17447018